CLINICAL TRIAL: NCT02015091
Title: VRC 314: A Phase 1, Open-Label, Clinical Trial With Experimental Controlled Human Malaria Infections (CHMI) to Evaluate Safety and Durability of Protection Following Intravenous and Intramuscular Administration of PFSPZ Vaccine in Malaria-Naive Adults
Brief Title: Study of Controlled Human Malaria Infections to Evaluate Protection After Intravenous or Intramuscular Administration of PfSPZ Vaccine in Malaria-Naive Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 140035; 14-I-0035
Record Dates: First submitted 2013-12-18; First posted 2013-12-19 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-09-08

CONDITIONS: Malaria
Keywords: Healthy Subjects; Vaccine-Mediated Protection; Immunogenicity; Sporozoites; Parasitemia
MeSH Terms: conditions — Malaria; Parasitemia

ARMS (4):
- 1, 4, 5, 6, 7 (Experimental): Vaccination schedules with 3 to 4 IV vaccinations per subject. Evaluation of protection against controlled human malaria infection (CHMI) is included.
  Interventions: Biological: PfSPZ Vaccine
- 2 (Experimental): Vaccination schedules 4 IM vaccinations per subject. Evaluation of protection against controlled human malaria infection (CHMI) is included.
  Interventions: Biological: PfSPZ Vaccine
- 3 (Experimental): Vaccination schedules 5 IV vaccinations per subject. Evaluation of protection against controlled human malaria infection (CHMI) is included.
  Interventions: Biological: PfSPZ Vaccine
- 8 (No Intervention): Participation in controlled human malari infection (CHMI) without prior vaccinations to serve as controls.

INTERVENTIONS:
Biological: PfSPZ Vaccine — The PfSPZ Vaccine is composed of radiation-attenuated Plasmodium falciparum sporozoites (PfSPZ) and is designed to prevent malaria in adults, children, and infants. It is formulated in phosphate buffered saline (PBS) with 1% human serum albumin (HSA). Sanaria Incorporated (Sanaria), Rockville, Maryland, developed and produced the PfSPZ Vaccine.
  Arms: 1, 4, 5, 6, 7; 2; 3

SUMMARY:
Background:

- People bitten by mosquitoes carrying weakened malaria parasites could fight off the disease if later exposed to normal malaria parasites. Scientists have discovered how to make the weakened parasites, which can be injected by the PfSPZ vaccine. Researchers want to see if people who receive the vaccine get malaria after being bitten in a controlled setting (a controlled human malaria infection, CHMI).

Objective:

- To see if the PfSPZ malaria vaccine is safe and prevents malaria in a controlled setting.

Eligibility:

- Healthy adults 18 45 years old.

Design:

* Participants will be screened with medical history, physical exam, blood and lab tests, and EKG.
* Participants will be split into 8 groups, to be in the study for 3 12 months.
* Participants will receive 3 5 vaccinations, injected by a needle in an arm vein or muscle.
* Participants will keep a health diary and be contacted by phone.
* For CHMI, a cup with mosquitoes carrying malaria is applied to participants arm for 5 minutes. Five mosquitoes at a time are used, until 5 have bitten. Some groups will be exposed to malaria more than once.
* After CHMI, participants will visit the clinic very frequently (including daily visits for 12 days) for 28 days.
* Blood will be drawn at most visits, from 1 to 20 tubes. Physical exam and medical history may also be repeated
* Participants who develop malaria will be treated immediately at the clinic. Standard treatment takes 72 hours. Malaria symptoms may last up to 3 days.

DETAILED DESCRIPTION:
VRC 314 is designed as an open-label evaluation of the safety, tolerability, immunogenicity and protective efficacy of PfSPZ Vaccine. This vaccine administered at 1.35 times 10(5) PfSPZ per injection by the IV route on a schedule of 5 vaccinations was previously shown to confer protection in all vaccinated subjects against CHMI performed shortly after last vaccination; however there was limited durability of protection in a small number of protected subjects who were rechallenged several months later. This study is designed to substantiate the initial results with the IV vaccination route for protection against CHMI. Based on the potential importance of dose and schedule in optimizing sustained immunity with this vaccine, an increase in PfSPZ IV dosage on schedules of 3 to 5 vaccinations will be evaluated for protection against CHMI conducted early (about 3 weeks) and late (about 24 weeks) after completion of vaccinations. To assess if a higher dose given by another route confers protection, one group will receive PfSPZ IM, with half of the amount administered in each arm on a schedule with 4 vaccination.

The primary objectives of the study are related to the safety and tolerability of vaccinations by the IV and IM routes of administration and protection against Plasmodium falciparum (Pf) challenge performed via a well-established CHMI procedure early (2-4 weeks) after completing schedules of 3 to 5 vaccinations. The secondary objective is related to the durability of protection at 20-26 weeks after the last vaccination and exploratory objectives are related to the immunogenicity of the PfSPZ Vaccine and identifying potential immune correlates of protection.

ELIGIBILITY:
* INCLUSION CRITERIA:

A volunteer must meet all of the following criteria to be included:

1. 18 to 45 years old adults.
2. Able and willing to participate for the duration of the study.
3. Able to provide proof of identity to the satisfaction of the study clinician completing the enrollment process.
4. Able and willing to complete the informed consent process.
5. Willing to donate blood for sample storage to be used for future research.
6. Willing to refrain from blood donation to blood banks for 3 years following P. falciparum CHMI.
7. Agrees not to travel to a malaria endemic region during the entire course of study participation.
8. Physical examination and laboratory results without clinically significant findings and a body mass index (BMI) less than or equal to 35 for vaccine groups or BMI less than or equal to 40 for control groups.
9. If enrolling into a Group with an IV vaccination schedule, then the physical exam must include assessment that there is adequate bilateral antecubital fossa venous access.

   Laboratory Criteria within 56 days prior to enrollment:
10. Hemoglobin greater than or equal to 11.2 g/dL for women; greater than or equal to 12.6 g/dL for men.
11. Differential and platelet count either within institutional normal range or accompanied by site physician approval.
12. Alanine aminotransferase (ALT) less than or equal to 1.25 x upper limit of normal (ULN) for vaccine groups or less than or equal to 1.75 x ULN for CHMI control groups.
13. Serum creatinine less than or equal to upper limit of normal.
14. Negative for HIV infection.

    Laboratory Criterion documented any time prior to enrollment:
15. Negative sickle cell screening test.

    Female-Specific Criteria:
16. Negative Beta-HCG pregnancy test (urine or serum) on day of enrollment for women presumed to be of childbearing potential.
17. A woman of childbearing potential must agree to use an effective means of birth control throughout the duration of study participation.

EXCLUSION CRITERIA:

A volunteer will be excluded if one or more of the following conditions apply:

1. Woman who is breast-feeding or planning to become pregnant during the time interval needed to complete the study.
2. Receipt of a malaria vaccine in a prior clinical trial.
3. Any history of malaria infection.
4. Evidence of increased cardiovascular disease risk; defined as >10% five year risk by the non-laboratory method.
5. Current use of systemic immunosuppressant pharmacotherapy.
6. History of a splenectomy, sickle cell disease or sickle cell trait.
7. Plan for major surgery between enrollment and challenge.
8. Known allergy to any component of the vaccine formulation; history of anaphylactic response to mosquito-bites; or known allergy to chloroquine phosphate, atovaquone or proguanil.
9. Participation in any study involving another investigational vaccine or drug within 12 weeks prior to enrollment, or plan to participate in another investigational vaccine/drug research during the study.
10. Personal beliefs that prohibit the receiving of vaccine product containing human serum albumin within the diluent.
11. Use or planned use of any drug with anti-malarial activity that would coincide with study vaccination or challenge.
12. History of psoriasis or porphyria, which may be exacerbated after treatment with chloroquine.
13. Anticipated use of medications known to cause drug reactions with chloroquine or atovaquone-proguanil (Malarone) such as cimetidine, metoclopramide, antacids, and kaolin.
14. Psychiatric condition that precludes compliance with the protocol; past or present psychoses; disorder requiring lithium; or within five years prior to enrollment, history of a suicide plan or attempt.
15. Any medical, psychiatric, social condition, occupational reason or other responsibility that, in the judgment of the investigator, is a contraindication to protocol participation or impairs a volunteer s ability to give informed consent or to comply with the protocol schedule.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 141 (Actual)
Dates: Start 2013-12-12; Primary Completion 2015-05-01 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of the metabolicallyactive,non-replicating, Plasmodium falciparum sporozoite (PfSPZ) vaccine (PfSPZ Vaccine) in malaria-naive healthy adults following multiple-dose IV administration. | The period of follow-up for each vaccinated subject is through at least 24 weeks after the last vaccination.
To evaluate the safety and tolerability of the metabolicallyactive,non-replicating, Plasmodium falciparum sporozoite(PfSPZ) vaccine (PfSPZ Vaccine) in malaria-naive healthyadults following multiple-dose IM administration. | The period of follow-up for each vaccinated subject is through at least 24 weeks after the last vaccination.
To determine if there is PfSPZ Vaccine-mediated protectionagainst infectious P. falciparum CHMI when the vaccine isadministered at 2.7 x 105 PfSPZ per injection by the IV routeusing a multi-dose schedule and the CHMI is administered at@... | At 4 weeks after CHMI.

SECONDARY OUTCOMES:
To determine if there is durability of PfSPZ Vaccine-mediatedprotection against infectious P. falciparum CHMI when the vaccine isadministered at 2.7 x 105 PfSPZ per injection by the IV route using amulti-dose schedule and the CHMI is ad... | At 4 weeks after CHMI.
To determine if there is PfSPZ Vaccine-mediated protection againstinfectious P. falciparum CHMI when the vaccine is administered at 2.2x 106 PfSPZ per injection by the IM route using a multi-dose schedule and the CHMI is administered at 2-... | At 4 weeks after CHMI.CHMI.
To determine if there is durability of PfSPZ Vaccine-mediatedprotection against infectious P. falciparum CHMI when the vaccine isadministered at 2.2 x 106 PfSPZ per injection by the IM route using a multi-dose schedule and the CHMI is admi... | At 4 weeks after CHMI.CHMI.

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Ledgerwood, D.O., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (2):
- United States (2):
  - University of Maryland Center for Vaccine Dev, Baltimore, Baltimore, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland

REFERENCES:
- [Background] Nussenzweig RS, Vanderberg J, Most H, Orton C. Protective immunity produced by the injection of x-irradiated sporozoites of plasmodium berghei. Nature. 1967 Oct 14;216(5111):160-2. doi: 10.1038/216160a0. No abstract available. PMID 6057225
- [Background] Seder RA, Chang LJ, Enama ME, Zephir KL, Sarwar UN, Gordon IJ, Holman LA, James ER, Billingsley PF, Gunasekera A, Richman A, Chakravarty S, Manoj A, Velmurugan S, Li M, Ruben AJ, Li T, Eappen AG, Stafford RE, Plummer SH, Hendel CS, Novik L, Costner PJ, Mendoza FH, Saunders JG, Nason MC, Richardson JH, Murphy J, Davidson SA, Richie TL, Sedegah M, Sutamihardja A, Fahle GA, Lyke KE, Laurens MB, Roederer M, Tewari K, Epstein JE, Sim BK, Ledgerwood JE, Graham BS, Hoffman SL; VRC 312 Study Team. Protection against malaria by intravenous immunization with a nonreplicating sporozoite vaccine. Science. 2013 Sep 20;341(6152):1359-65. doi: 10.1126/science.1241800. Epub 2013 Aug 8. PMID 23929949
- [Background] Epstein JE, Tewari K, Lyke KE, Sim BK, Billingsley PF, Laurens MB, Gunasekera A, Chakravarty S, James ER, Sedegah M, Richman A, Velmurugan S, Reyes S, Li M, Tucker K, Ahumada A, Ruben AJ, Li T, Stafford R, Eappen AG, Tamminga C, Bennett JW, Ockenhouse CF, Murphy JR, Komisar J, Thomas N, Loyevsky M, Birkett A, Plowe CV, Loucq C, Edelman R, Richie TL, Seder RA, Hoffman SL. Live attenuated malaria vaccine designed to protect through hepatic CD8(+) T cell immunity. Science. 2011 Oct 28;334(6055):475-80. doi: 10.1126/science.1211548. Epub 2011 Sep 8. PMID 21903775